CLINICAL TRIAL: NCT00437528
Title: Phase I Study for Evaluating the Safety and Applicability of a Novel Heat Flow Sensor Unit for Measuring Urinary Bladder Capacity
Brief Title: Safety and Applicability Study of a Novel Heat Flow Sensor Unit for Measuring Urinary Bladder Capacity
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rambam Health Care Campus (Other)
Other Study IDs: 2456_CTIL
Record Dates: First submitted 2007-02-19; First posted 2007-02-21 (Estimated); Last update posted 2007-05-17 (Estimated); Status verified 2007-02

CONDITIONS: Overactive Bladder; Urge Urinary Incontinence; Enuresis; Self Clean Intermittent Catheterization
Keywords: Heat flow; Sensor; Overactive bladder; Urinary incontinence
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence, Urge; Enuresis; Urinary Incontinence

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
A novel sensor (a device named sensurine)was developed in the aim of real- time measurement of bladder volume. The sensurine device is a wearable, fully passive, non-invasive and compact heat flow sensor (patent pending) and electronic control unit. The device will serve as a tool for managing and treating bladder dysfunction (by behavioral treatment), such as overactive bladder without incontinence, urge incontinence and voiding difficulties. In this phase I of the clinical trial the sensor unit will be tested for technological feasibility demonstration and for collecting design data.

DETAILED DESCRIPTION:
The Primary objectives are to asses the safety and the physical performance of the SenseUrine's sensor unit and to validate the concept of determining bladder volume by measuring heat flow. The Secondary objective is to optimize the device accuracy Primary endpoints: To show that the sensor has no negative effect on the subject, to determine bladder urine volume, based on the sensor's signals, in an accuracy of ±10% compared to the actual volume. Secondary endpoint - to determine bladder urine volume, in an accuracy of ±10%, in different ambient conditions (temperature and clothing).

Inclusion criteria - All subjects will be aged 18-50, active, in good general health and without urinary complaints or documented urinary tract dysfunctions. Exclusion criteria - Pregnancy, breast feeding, known allergic sensitivity to medical adhesive tapes, cognitive incompatibility and mental incompetence.

On the first visit, the subject will sign an informed consent form. A medical intake including demographic data will be collected. Stage 1 will serve for basic testing of the sensor unit and for measuring the maximal and minimal bladder volume. The sensor will be attached to the lower abdomen wall and checked for functionality. Each subject will fill up his bladder (by drinking water) until sensing a strong urge to void. The subject will then void until he is empty into a measurement cup. Ultrasound measurement (US) of bladder volume, and sensor signal will be read and recorded by a standard miliVoltmeter just before and immediately after emptying the bladder. Sensor, US and cup measurement readings will not be done by the same investigator. Continuing to stage 2 will depend on the preliminary results (sensor readings compared to the measured volume and US readings) determining feasibility.. Stage 2 will serve for measuring the dynamics of bladder heat conductivity during the filling and voiding phases. On the 2nd visit the subject will fill up his bladder by gradually drinking 500CC of water (over 60-90 minutes) until sensing a strong urge to void. The subject will drink an additional 50-100CC of water and wait around 10 minutes in the aim of achieving maximal bladder capacity. The sensor signals will be recorded from the beginning of this bladder filling stage every 5-10 minutes. Then, the subject will be requested to void in a controlled manner and to intentionally stop urinating after emptying 50-100CC of urine (voided volume will be determined by the measurement cup). The controlled voiding of 50-100CC will be repeated until the bladder is empty. The sensor signals will be read and recorded during both stages. Visit 3 will be performed in the same manner but in different positions during measurements (supine-on the back, sides and front, sitting, and standing). Visit 4 (final visit) will serve for demonstrating the sensor unit's performance in different ambient temperature and clothing. Two subjects will be randomly selected to examine the sensor in an ambient of 15ºC (this will be controlled by an air-conditioned room with an external thermometer) for measuring the dynamic range (maximal and minimal bladder capacity). The same will be done at room temperature twice- with light and heavy clothing. The other 2 subjects will be randomly selected to examine the sensor's performance in an ambient of 40ºC (hot temperature will be achieved by an electric heater in a small room controlled with an external thermometer) for measuring the dynamic range (maximal and minimal bladder capacity). The same will be done at room temperature twice- with light and heavy clothing.

All output signals will be logged and processed to show the correlation between the calculated heat conductance of the bladder and the volume. A table consisting the calculated indexes of conductivity vs. bladder volumes will be designed.

General: 10 subjects will be recruited by advertisement with notification of some compensation for their time and travel to the study site. Every session will last about 4 hours long. In each working day 3-5 subjects will participate and the total trial period is expected to be approximately 20 working days.

ELIGIBILITY:
Inclusion Criteria:

* All subjects will be aged 18-50, active, in good general health and without urinary complaints or documented urinary tract dysfunctions

Exclusion Criteria:

* Pregnancy, breast feeding, known allergic sensitivity to medical adhesive tapes, cognitive incompatibility and mental incompetence

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2006-11; Study Completion 2007-12

CONTACTS AND LOCATIONS:
Overall Officials: Yoram Vardi, Prof, Principal Investigator — Rambam Health Campus; Ilan Gruenwald, MD, Study Director — Rambam Health Campus; Irena Papier, RN, MPA, Study Director — Rambam Health Campus
Locations (1):
- Rambam Healthcare Campus, Haifa, Northern District, Israel